CLINICAL TRIAL: NCT04029714
Title: A Multicentre Randomised Active Surveillance (AS) Trial of Current Practice Versus Standardised Triggers for Curative Treatment of Prostate Cancer
Brief Title: Prostate Cancer Active Surveillance Trigger Trial (PCASTT-UK): Comparing Current Practice for Men With Prostate Cancer on Active Surveillance (AS) to an AS Protocol With Standardised Triggers for Transitioning to Curative Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: King's College London (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 228445
Record Dates: First submitted 2019-07-16; First posted 2019-07-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Active Surveillance; MRI; standardised treatment triggers; randomized
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Current practice for active surveillance (Active Comparator): In this arm, patients are monitored according to current practice for active surveillance at the trial centre. Repeat biopsies (and/or other examinations) and initiation of curative treatment are performed according to the urologist's judgement.
  Interventions: Procedure: Active Surveillance
- Arm 2: Standardized triggers for treatment (Experimental): In this arm, patients are monitored according to a standardized active surveillance protocol with specific triggers for treatment. Repeat biopsies and curative treatment are only initiated if/when specific criteria are fulfilled.
  Interventions: Procedure: Active Surveillance

INTERVENTIONS:
Procedure: Active Surveillance — Active monitoring of prostate cancer and curative treatment if there are signs of tumor progression.

SUMMARY:
A large proportion of men with prostate cancer are overdiagnosed and overtreated mainly due to PSA testing. Active surveillance (AS) aims to reduce these harms by recommending curative treatment only when and if signs of tumour progression occur. There are however a number of uncertainties in AS, the most important being when to initiate treatment.

Therefore, the Scandinavian Prostate Cancer Group (SPCG) are running a large multi-centre randomised control trial (RCT) to test the safety of a standardized active surveillance protocol with specific triggers for repeat biopsies and initiation of curative treatment, compared to the current practice for active surveillance. They are recruiting in multiple sites in Sweden, Denmark and Finland. The primary aim is to reduce overtreatment and subsequent side effects, without increasing the risk of disease progression or prostate cancer mortality.

In the UK, there is also no set criteria for when to re-biopsy and/or initiate curative treatment for patients on AS and tends to be at the clinician's discretion. Thus, PCASTT-UK has been established to run as a parallel RCT and add to the findings from SPCG-17.

DETAILED DESCRIPTION:
STUDY HYPOTHESIS The aim of this trial is to test the safety of an Active Surveillance protocol comparing current practice to standardized triggers for initiation of curative treatment, based on Magnetic Resonance Imaging or biopsy pathology. The study hypothesis is that standardized triggers will reduce overtreatment without increasing disease progression and prostate cancer mortality.

STUDY DESIGN Randomized multi-centre open-label clinical trial.

INTERVENTIONS Patients within 12 months of a diagnosis of prostate cancer will be approached and consented to the study. Computerised randomisation (1:1) will assign participants to either the control (Arm 1) or intervention arm (Arm 2). In the control arm, patients will be treated according to active surveillance protocol at the trial centre; in the intervention arm patients will follow standardised active surveillance protocol applying specific criteria for repeat biopsies and the initiation of curative treatment. Patients are stratified by centre and Gleason score.

FOLLOW UP In both arms, patients will followed up for 10 years with the following schedule: a PSA test every 6 months, clinical examination (with PSA test) and Quality of Life (QoL) questionnaire annually, and MRI every second year. Re-biopsy and/or initiation of curative treatment depends on the trial arm patients are randomised to.

Repeat biopsies

Arm 1 (control arm): according to current practice (urologists' judgement)

Arm 2 (intervention arm): standardised triggers

* A systematic repeat biopsy if PSA density increases to > 0.2 ng/ml/cc, and then at every 0.1 ng/ml/cc increase
* MRI progression in men with previously only Gleason grade 3+3: 5 mm or more increase in size in any dimension of a measurable lesion, increase in PI-RADS score to 3-5, a new lesion with PI-RADS score 3-5, or high or very high suspicion of extra-capsular extension or seminal vesicle invasion
* MRI progression in men with Gleason grade 3+4: 5 mm or more increase in size in any dimension of a measurable lesion, or a new lesion with PI-RADS score 3-5

Curative treatment

Arm 1 (control arm): According to current practice (urologists judgement)

Arm 2 (intervention arm): standardised triggers

* MRI progression in lesions with confirmed Gleason grade 4: increase in PI-RADS score to 4 or 5, or high or very high suspicion of extra-capsular extension or seminal vesicle invasion
* Pathological progression: Gleason pattern 5, primary Gleason pattern 4 in any core with 5 mm or more cancer, Gleason 3+4 in 3 or more cores or 30% if more than 10 cores are taken, or Gleason 3+4 in 10 mm or more cancer

Patients will remain on trial unless they end Active Surveillance due to initiation of treatment, development of metastases, transition to watchful waiting, or death of any cause. After the initiation of curative treatment, watchful waiting, or palliative treatment for cancer progression, the patient is treated according to the standard protocol of the participating centre.

ELIGIBILITY:
Inclusion Criteria:

* Recently (within 12 months) diagnosed adenocarcinoma of the prostate
* Tumour stage ≤ T2a, NX, M0 (former MX)
* PSA <15ng/ml, PSA density ≤ 0.2 ng/ml/cm3
* Gleason pattern 3+3=6 (any number of cores, any cancer involvement) or Gleason pattern 3+4=7 (<3 cores (or ≤30 % of cores if more than ten cores), <10 mm cancer in one core)
* Life expectancy >10 years with no upper age limit*
* Candidate for curative treatment if progression occurs
* Signed written informed consent.

  * There is no upper age limit; however the estimated remaining lifetime for the patient should be more than ten years. The potential life expectancy of the participants should be estimated based on age, co-morbidity and risk factors for death, such as frailty and smoking.

Exclusion Criteria:

* Not eligible for AS according to above criteria
* Not competent in spoken or written English

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2019-09-19 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Median 10 years follow-up
  Progression-free survival is defined as cumulative incidence of PSA relapse following curative treatment and cumulative incidence of androgen therapy in untreated men. Following radical prostatectomy, biochemical recurrence is defined by two consecutively rising PSA values >0.2 ng/ml. After radiotherapy (RT) with or without androgen deprivation therapy, the definition of PSA failure is any rise by 2 ng/ml or more above the nadir PSA value, regardless of the serum concentration of the nadir.

SECONDARY OUTCOMES:
Cumulative incidence of pT3 at radical prostatectomy specimens | Median 10 years follow-up
  Occurrence of confirmed pT3 in radical prostatectomy specimens according to the pathology report
Cumulative incidence of metastases | Median 10 years follow-up
  Occurrence of distant metastasis (suspected or confirmed) during follow-up
Cumulative number of treatments with curative intent (mainly radical prostatectomies or local radiotherapy) | Median 10 years follow-up
  Occurrence of radical prostatectomies or local radiotherapy (with or without adjuvant androgen deprivation therapy)
Cumulative incidence of switch to watchful waiting | Median 10 years follow-up
  Occurrence of conversions from active surveillance to watchful waiting during follow-up
Quality of life assessed by EPIC-26 score, incontinence, erectile dysfunction, self-reported quality of life: questionnaires | Median 10 years follow-up
  Assessed by questionnaires at baseline and every second year.
  Quality-of-life data will be presented as proportions with symptoms and relative risks. Outcome variables will be dichotomized using predetermined cut-off values.
  The following parameters will be included in the analysis:
  * EPIC-26 score
  * Incontinence
  * Erectile dysfunction
  * Self-reported quality of life (rated on a scale of 1-7)

CONTACTS AND LOCATIONS:
Locations (5):
- United Kingdom (5):
  - Bedford Hospital, Bedford
  - Epsom & St. Helier, London
  - Guy's Hospital, London
  - Queen Elizabeth Hospital, London
  - Royal Mardsen Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided